CLINICAL TRIAL: NCT04504110
Title: A Prospective Study to Evaluate 68Ga-FAPI-04 and 18F-FDG PET/CT in Patients With Epithelial Ovarian Cancer: Compared With Histological Findings
Brief Title: 68Ga-FAPI-04 and 18F-FDG PET/CT in Patients With Epithelial Ovarian Cancer: Compared With Histological Findings
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAPIEOC
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epithelial ovarian cancer (Experimental): 68Ga-FAPI-04 and 18F-FDG PET/CT
  Interventions: Diagnostic Test: 68Ga-FAPI-04 PET/CT and 18F-FDG PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI-04 PET/CT and 18F-FDG PET/CT — Patients with epithelial ovarian cancer who are scheduled for surgical intervention will undergo a comparative 68Ga-FAPI-04 and 18F-FDG PET/CT study before the surgery.

SUMMARY:
Epithelial ovarian cancer (EOC) is a tumor entity featured by frequent involvement of peritoneum, also called peritoneal carcinomatosis. It is a type of metastasis accompanied by significant cancer-associated fibroblasts (CAFs) accumulation. Fibroblast activation protein (FAP) is a protein that is overexpressed on CAFs and can be non-invasively monitored by a novel radiotracer called 68Ga-FAPI-04 positron emission tomography/computed tomography (PET/CT). In this study, we will explore the value of 68Ga-FAPI-04 PET/CT in patients with epithelial ovarian cancer who are scheduled for surgical intervention. The findings of 68Ga-FAPI-04 PET/CT will also be compared with that of 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (18F-FDG) PET/CT, which is one of the most commonly used modalities in evaluating EOC, and histological findings.

DETAILED DESCRIPTION:
Patients with epithelial ovarian cancer who are scheduled for surgical intervention will be recruited in this study. They will undergo a comparative 68Ga-FAPI-04 and 18F-FDG PET/CT study before the surgery. No tumor-specific treatment is allowed between the scan and surgery, e.g. adjuvant chemotherapy, neoadjuvant chemotherapy, and intraperitoneal chemotherapy. Three types of lesions will be marked based on 68Ga-FAPI-04 and 18F-FDG PET/CT findings, which is FAPI+/FDG-, FAPI-/FAPI+, and FAPI+/FDG+ lesions. The marked lesions will be explored by the surgeon, resected if possible, and compared with histological results. A fourth type of lesion will be added into the analysis if that lesion is both FAPI and FAP negative but is a histological-confirmed positive lesion.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed
* EOC patients who are scheduled for surgery. The diagnosis of EOC should be based on the previous histological results or cytological evaluation combined with a serum CA-125 to carcinoembryonic antigen ratio>25 to confirm the primary diagnosis and exclude a nongynecologic cancer.

Exclusion Criteria:

* Known hypersensitivity to any of the excipients of 18F-FDG and 68Ga-FAPI-04.
* Tumor-specific treatment is necessary between the scans and surgery, e.g. adjuvant chemotherapy, neoadjuvant chemotherapy, and intraperitoneal chemotherapy.
* Pregnant or breast-feeding women.
* Any mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the study, and/or evidence of an uncooperative attitude.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian cancer is a female-specific tumor entity.
Enrollment: 30 (Estimated)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
SUVmax of positive lesions | 1 hour after tracer injection
  68Ga-FAPI-04 and 18F-FDG accumulation will be determined using SUVmax

SECONDARY OUTCOMES:
Histological findings | 60 day after surgery
  The presence of tumor cells on resected specimen will be evaluated by pathologists. The FAP expression will be determined using immunohistochemical staining using anti-FAP antibody (Abcam).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No